CLINICAL TRIAL: NCT01237626
Title: The CIHR Team in Driving in Older Persons (Candrive II) Research Program
Brief Title: CIHR Team in Driving in Older Persons
Acronym: CANDRIVE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other); Lakehead University (Other); McGill University (Other); University of British Columbia (Other); University of Manitoba (Other); University of Waterloo (Other); University of Toronto (Other); University of Western Ontario, Canada (Other); University of Victoria (Other); McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: #2008610-01H
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Aging and Health and Impact on Driving
Keywords: Driving; Aging; Older drivers; Medical Fitness to drive; Health Status; At-fault collisions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The following study is designed in order to effectively collaborate and coordinate information amongst colleagues to advance knowledge on information related to older drivers. Candrive is dedicated to improving the safety and quality of life of older drivers. The major objective is to develop a valid, easy to use in office screening tool that will help clinicians identify older drivers who need further assessment of their driving. Over the course of the study, the goal will be to provide enough data to establish findings relating to knowledge generation, translation of research into action, training and sustainability. It is our hope that the research process will translate to help increase the knowledge of public policy makers, clinicians and the general public. A 5 year study will create an opportunity to document the natural course of an older adult's driving patterns up until driving cessation. This will not only provide data for road safety but also help understand the psychosocial factors leading to driving cessation. The data relating to psychosocial factors may also lead the way in establishing ways of extending the safe driving period for older adults.

The investigators hypothesize that the knowledge derived from this interdisciplinary research will be used by transportation policy makers, clinicians, and general public to improve safety and quality of life for older drivers.

DETAILED DESCRIPTION:
Driving a motor vehicle has become an everyday necessity in modern Canadian culture. The privilege of maintaining a valid driver's license promotes an independent lifestyle (Voelker, 1999). Since driving is a demanding task that requires a high level of mental and physical skills, it is critical that those who obtain a valid driver's license are medically fit to operate a motor vehicle. Adverse health conditions make driving difficult based on the high cognitive and physical demand (Man-Son-Hing, 2007, Marshall, 2008). The loss of driving privileges due to chronic health conditions can have a negative effect on an individual's quality of life. These individuals require greater community support and suffer from low self-esteem (Fonda, 2001, Ragland, 2004, Ansley et al., 2004). As much as it is desirable to promote independence, the safety implications of driving require careful consideration.

In Canada, persons over the age of 65 represent the fastest growing segment of the population. This age group is predicted to make up 24 % of the total population by the year 2030 (CMA Journal, 1994, Stats Can, 2005). As a result, the number of older persons holding a driver's license has increased in both percentage and absolute terms (Ont Road Safety, 2004, Transport Can, 2001, Ragland, 2004, Ansley et al., 2004). Therefore, it is not surprising that those over 70 years of age have the highest crash rates per mile driven (Brorsson, 1989, Stutts & Wilkins, 2003, Gresset & Meyer, 1994, Cotrell & Wild, 1999, Rizzo et al., 2001, Meddinger-Rapport, 2002, Ansley et al., 2004).

Candrive is an interdisciplinary health research program dedicated to improving the safety of older drivers in Canada. The members of Candrive believe that establishing a comprehensive approach to aging driver issues will reduce the morbidity and mortality associated with motor vehicle crashes and allow older Canadian drivers to maintain their independence and healthy lifestyles.

A major focus of the Canadian Institutes of Health Research (CIHR) Team Grant is to conduct the Common Cohort study, a study in which 1000 drivers age 70 or older will be recruited and followed for 5 years. The Common Cohort study involves 7 sites (Victoria, Winnipeg, Thunder Bay, Hamilton, Toronto, Ottawa, and Montreal) in 4 provinces. Participants in the Common Cohort study will undergo comprehensive annual assessments as well as having their driving patterns monitored for 5 years. One of the major objectives of the Common Cohort study will be the development of a valid, easy-to-use in-office screening tool that will help clinicians identify older drivers who may need further assessment of their driving ability.

The vision of Candrive is to use a national interdisciplinary research approach to improve the safety and health-related quality-of-life of older drivers. Collaboration with key stakeholders throughout the process ensures that research products will translate into public policy and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. have a general class driver's license and actively driving for at least 1 year
2. have vehicle access
3. drive at least 4 times a week (4 round trips)
4. reside in the local regions of one of the study cities (Victoria, Winnipeg, Thunder Bay, Ottawa, Toronto, Hamilton or Montreal)
5. consent to release driving information from the provincial Ministry of Transportation
6. agree to undergo annual physical and cognitive assessment and be contacted at least quarterly for data pick up and interview
7. be under the care of a family physician
8. have a primary vehicle for driving that is model year 1996 or newer
9. be age 70 or greater
10. have a life expectancy of at least 5 years
11. be fluent in either French or English
12. drive one vehicle 70% of the time or greater
13. reside in the province at least 10 months of the year.

Exclusion Criteria:

1. moved out of the province
2. contradiction to driving, within the last 6 months, according to the Canadian Medical Association Guidelines (7th edition), such as heart attack or low blood sugar
3. diagnosis of a progressive condition, such as dementia, Alzheimer's disease, and/or macular degeneration.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The cohort will be established in 7 cities in 4 provinces, including Ontario (Ottawa, Thunder Bay, Toronto, Hamilton), Quebec (Montreal), Manitoba (Winnipeg) and British Columbia (Victoria). Participants will be recruited through the media - newspapers (community and city), radio, public presentations and newsletters to senior associations. We have established collaboration with two senior organizations; Canada's Association for the Fifty-plus (CARP) and the Federal Superannuates National Association (FSNA). These senior organizations will be targeted through mail out letters and presentations at annual meetings. Additionally, recruitment posters will be displayed at local community centres, fitness centres, doctor's offices, hospitals and other clinic waiting rooms.
Sampling Method: Non-Probability Sample
Enrollment: 932 (Actual)
Dates: Start 2008-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
At-Fault Motor Vehicle Collisions (MVC) | Throughout the 5-year period
  Motor Vehicle Collision as determined through the provincial Ministry of Transportation records.

SECONDARY OUTCOMES:
Health Status | Any point throughout 5-year study
  Physical, cognitive (i.e. Montreal Cognitive Assessment) and psychological assessment measures

CONTACTS AND LOCATIONS:
Overall Officials: Shawn C Marshall, MD MSc FRCPC, Principal Investigator — The Ottawa Hospital Research Institute; Malcom Man-Son-Hing, MD, Principal Investigator — The Ottawa Hospital Research Institute
Locations (7):
- Canada (7):
  - University of Victoria, Victoria, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Lakehead University, Thunder Bay, Ontario
  - Toronto Rehabilitation Institue, Toronto, Ontario
  - School of Physical and Occupational Therapy McGill University, Montreal, Quebec

REFERENCES:
- [Background] Eby DW, Molnar LJ. Driving fitness and cognitive impairment: issues for physicians. JAMA. 2010 Apr 28;303(16):1642-3. doi: 10.1001/jama.2010.495. No abstract available. PMID 20424255
- [Background] Caragata, G.E., Tuokko, H., & Damini, A. (2009). Fit to Drive: A Pilot Study to Improve the Physical Fitness of Older Drivers. Activities, Adaptation & Aging, 33(4), 240-255.
- [Background] Marshall SC. The role of reduced fitness to drive due to medical impairments in explaining crashes involving older drivers. Traffic Inj Prev. 2008 Aug;9(4):291-8. doi: 10.1080/15389580801895244. PMID 18696384
- [Background] Dickerson AE, Molnar LJ, Eby DW, Adler G, Bedard M, Berg-Weger M, Classen S, Foley D, Horowitz A, Kerschner H, Page O, Silverstein NM, Staplin L, Trujillo L. Transportation and aging: a research agenda for advancing safe mobility. Gerontologist. 2007 Oct;47(5):578-90. doi: 10.1093/geront/47.5.578. PMID 17989400
- [Background] Tuokko HA, Rhodes RE, Dean R. Health conditions, health symptoms and driving difficulties in older adults. Age Ageing. 2007 Jul;36(4):389-94. doi: 10.1093/ageing/afm032. Epub 2007 Mar 24. PMID 17384420
- [Background] Man-Son-Hing M, Marshall SC, Molnar FJ, Wilson KG. Systematic review of driving risk and the efficacy of compensatory strategies in persons with dementia. J Am Geriatr Soc. 2007 Jun;55(6):878-84. doi: 10.1111/j.1532-5415.2007.01177.x. PMID 17537088
- [Background] Marshall SC, Wilson KG, Molnar FJ, Man-Son-Hing M, Stiell I, Porter MM. Measurement of driving patterns of older adults using data logging devices with and without global positioning system capability. Traffic Inj Prev. 2007 Sep;8(3):260-6. doi: 10.1080/15389580701281792. PMID 17710716
- [Derived] Rapoport MJ, Naglie G, Weegar K, Myers A, Cameron D, Crizzle A, Korner-Bitensky N, Tuokko H, Vrkljan B, Bedard M, Porter MM, Mazer B, Gelinas I, Man-Son-Hing M, Marshall S. The relationship between cognitive performance, perceptions of driving comfort and abilities, and self-reported driving restrictions among healthy older drivers. Accid Anal Prev. 2013 Dec;61:288-95. doi: 10.1016/j.aap.2013.03.030. Epub 2013 Mar 30. PMID 23601097
- [Derived] Marshall SC, Man-Son-Hing M, Bedard M, Charlton J, Gagnon S, Gelinas I, Koppel S, Korner-Bitensky N, Langford J, Mazer B, Myers A, Naglie G, Polgar J, Porter MM, Rapoport M, Tuokko H, Vrkljan B, Woolnough A. Protocol for Candrive II/Ozcandrive, a multicentre prospective older driver cohort study. Accid Anal Prev. 2013 Dec;61:245-52. doi: 10.1016/j.aap.2013.02.009. Epub 2013 Mar 7. PMID 23541299
- [Derived] Smith A, Marshall S, Porter M, Ha L, Bedard M, Gelinas I, Man-Son-Hing M, Mazer B, Rapoport M, Tuokko H, Vrkljan B. Stability of physical assessment of older drivers over 1 year. Accid Anal Prev. 2013 Dec;61:261-6. doi: 10.1016/j.aap.2013.02.007. Epub 2013 Feb 13. PMID 23489912
- See also: Candrive website — http://www.candrive.ca